CLINICAL TRIAL: NCT00002338
Title: A Phase I Trial to Evaluate the Safety, Tolerance, and Pharmacokinetics of 935U83 After Multiple Dosing in Patients With HIV Infection
Brief Title: The Safety and Effectiveness of 935U83 in HIV-Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 237A; 02
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-04

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — raluridine

INTERVENTIONS:
Drug: Raluridine

SUMMARY:
To assess the safety, tolerance, and steady-state pharmacokinetics of multiple oral doses of 935U83 administered to patients with HIV infection. To obtain preliminary evidence of antiretroviral activity of 935U83. To prospectively evaluate the emergence of in vitro drug resistance. To determine the effects of 935U83 dosing on CD4+ cell counts.

DETAILED DESCRIPTION:
Patients (10 per dose level) are randomized to receive 1 of 4 doses of 935U83 every 8 hours for 12 weeks. Five patients at each dose level must complete 4 weeks of treatment without serious toxicity before subsequent patients are entered at the next higher dose. If lack of antiretroviral effect or unacceptable toxicity is demonstrated at a particular dose level, the dose regimens may be adjusted.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Recommended:

* PCP prophylaxis for patients whose CD4 counts fall below 200 cells/mm3 or who develop PCP during study participation.

Allowed:

* Acute treatment and secondary prophylaxis for tuberculosis, Mycobacterium avium intracellulare, toxoplasmosis, histoplasmosis, cryptococcosis, disseminated candidiasis, or cytomegalovirus infection.

Patients must have:

* HIV infection.
* CD4 count 200 - 500 cells/mm3.
* No history of or current AIDS-defining indicator disease by CDC criteria.
* No antiretroviral therapy within the past 6 months.
* Consent of parent or guardian if less than 18 years of age.

Exclusion Criteria

Co-existing Condition:

Patient with the following symptoms or conditions are excluded:

* Current evidence of chronic hepatitis of any etiology.
* Seropositivity for HBsAg or hepatitis C virus by second generation ELISA.

Concurrent Medication:

Excluded:

* Cytotoxic chemotherapy.
* Other antiretroviral drugs.
* Immunomodulators.
* Foscarnet.
* GM-CSF or G-CSF.
* Erythropoietin.

Concurrent Treatment:

Excluded:

* Radiation therapy.

Patients with the following prior conditions are excluded:

History of chemical, viral, or alcohol-induced clinical hepatitis within the past 3 years.

Prior Medication:

Excluded within the past 6 months:

* Any antiretroviral therapy.
* HIV immunotherapeutic vaccine.

Excluded within the past 4 weeks:

* Cytotoxic chemotherapy.
* Immunomodulating agents such as systemic corticosteroids, IL-2, alpha interferon, beta interferon, or gamma interferon.

Prior Treatment:

Excluded within the past 4 weeks:

* Radiation therapy. Current alcohol or illicit drug use that may interfere with study compliance.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - ViRx Inc, San Francisco, California
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Goodgame Med Group, Maitland, Florida
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Duke Univ Med Ctr, Durham, North Carolina
  - Univ of Cincinnati / Holmes Hosp, Cincinnati, Ohio
  - Univ of Pittsburgh Med School, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Riddler SA, Wang LH, Bartlett JA, Savina PM, Packard MV, McMahon DK, Blum MR, Dunn JA, Elkins MM, Mellors JW. Safety and pharmacokinetics of 5-chloro-2',3'-dideoxy-3'-fluorouridine (935U83) following oral administration of escalating single doses in human immunodeficiency virus-infected adults. Antimicrob Agents Chemother. 1996 Dec;40(12):2842-7. doi: 10.1128/AAC.40.12.2842. PMID 9124852